CLINICAL TRIAL: NCT03726645
Title: The Role of Gut Microbiota in the Pathogenesis of Ankylosing Spondylitis (AS), and the Effect of Fecal Microbiota Transplantation on Gut Microbiota, Gut Wall Inflammation and Clinical Activity of AS
Brief Title: The Effect of Fecal Microbiota Transplantation in Ankylosing Spondylitis (AS) Patients.
Acronym: ASGUT
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hospital District of Helsinki and Uusimaa (Other)
Responsible Party: Principal Investigator, Johanna Hiltunen, MD, Principal Investigator, Hospital District of Helsinki and Uusimaa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HospitalDHU/Rheumatology
Record Dates: First submitted 2018-03-23; First posted 2018-10-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Ankylosing Spondylitis
Keywords: ankylosing spondylitis; fecal microbiota transplantation; intestinal mucosal immunity; dysbiosis; microbiome
MeSH Terms: conditions — Spondylitis, Ankylosing; Dysbiosis | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: FMT type (donor/own feces) randomization is done by a study nurse.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): Allogeneic fecal microbiota transplantation (from donor)
  Interventions: Other: Fecal microbiota transplantation
- Control group (Placebo Comparator): Autologous fecal microbiota transplantation (own stool)
  Interventions: Other: Fecal microbiota transplantation

INTERVENTIONS:
Other: Fecal microbiota transplantation — Fecal microbiota transplantation

SUMMARY:
Ankylosing spondylitis (AS) patients often have subclinical gut wall inflammation. Gut dysbiosis has been associated with both AS and Crohn disease, both of which have several features in common. Gut dysbiosis is associated with specific microbial profile in AS patients. Fecal microbiota transplantation (FMT) has been proved to be safe and effective treatment for recurrent Clostridium difficile infection, and the change in gut microbiota is shown to be long lasting. It has led to interest to study its effect on different inflammatory conditions associated with gut dysbiosis.

We hypothesize that dysbiosis in AS leads to inflammasome overactivation on gut mucosa. We aim to study the role of gut inflammation, gut microbiota and inflammasome activation in pathogenesis of AS, and the effect of FMT on these factors, as well as clinical activity, in AS patients.

DETAILED DESCRIPTION:
This is a double-blind placebo- controlled randomized pilot study with 20 patients with active AS from 2 Finnish outpatient clinics. An ileocolonoscopy will be performed to all patients. 10 patients will receive FMT with feces of one of two healthy donors, and 10 patients with their own feces during ileocolonoscopy. Ileal and colonic biopsies will be taken to assess gut wall inflammation and mucosal microbiota composition. Ileocolonoscopy will be controlled in 6 months in patients with macroscopic inflammatory lesions in the first colonoscopy. From mucosal biopsies we will assess intestinal mucosal structure, inflammasome activity, cytokine expression, and the mucin layer thickness and the amount of bacterial LPS (lipopolysaccharide), which are associated with mucosal integrity. Blood levels of zonulin and LPS as indicators of mucosal permeability and bacterial penetrance will be assessed. Fecal samples will be collected repeatedly to measure fecal calprotectin, and to assess the bacterial profile changes. From mucosal biopsies and fecal samples microbial DNA will be segregated and bacterial species sorted by rRNA- based sequence technique. Clinical activity of AS will be assessed in follow-up visits as well as repeated BASDAI (Bath Ankylosing Spondylitis Disease Activity Index), BASFI (Bath Ankylosing Spondylitis Functional Index) and MASES (Maastricht Ankylosing Spondylitis Enthesitis Score) evaluations, and measurement of CRP (C-reactive protein) and ESR (erythrocyte sedimentation rate). Follow-up time is 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AS by either the 1984 New York criteria or the ASAS (Assessment of SpondyloArthritis International Society) criteria for axial spondyloarthritis.
* Active disease measured by BASDAI > 4.
* Availability of consecutive fecal samples over 1 year period.
* Compliance to attend ileocolonoscopy and FMT procedure.

Exclusion Criteria:

* Diagnosis of inflammatory bowel disease.
* Antibiotic therapy within the last 3 months.
* Use of any probiotics within the last 3 months.
* Pregnancy.
* Unability to provide a written consent.
* Other reason which by the opinion of the investigator makes patient ineligible for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
The effect of FMT (fecal microbiota transplantation) on the clinical activity of ankylosing spondylitis (AS) as assessed by change in BASDAI (Bath Ankylosing Spondylitis Disease Activity Index). | 5 measurements within 12 months
  BASDAI scale 0-10 (the higher the score the more severe the symptoms). Decrease in BASDAI indicates positive outcome.

SECONDARY OUTCOMES:
The effect of FMT on the clinical activity of AS as assessed by change in BASFI (Bath Ankylosing Spondylitis Functional Index). | 5 measurements within 12 months.
  BASFI scale 0-10 (the higher the score the more severe the symptoms). Decrease in BASFI indicates positive outcome.
The effect of FMT on the clinical activity of AS as assessed by change in MASES (Maastricht Ankylosing Spondylitis Enthesitis Score). | 5 measurements within 12 months.
  MASES scale 0-13 (the higher the score the more severe the symptoms). Decrease in MASES indicates positive outcome.
The effect of FMT on C-reactive protein (CRP) concentration. | 7 measurements within 12 months.
  Change in inflammatory parameter CRP concentration indicates positive outcome.
The effect of FMT on erythrocyte sedimentation rate (ESR) level. | 7 measurements within 12 months.
  Change in inflammatory parameter ESR level indicates positive outcome.
The effect of FMT on gut wall inflammation as assessed by change in fecal calprotectin (F-calpro) level. | 7 measurements within 12 months.
  Change in fecal calprotectin level indicates positive outcome.
The effect of FMT on gut microbiota composition in AS patients. | 7 stool microbial analysis within 12 months.
  Change in gut microbiota composition evaluated by stool microbial analysis indicates positive outcome.
Association between specific intestinal pathogens and disease activity as assessed by BASDAI score. | 7 stool microbial samples and 5 BASDAI measurements within 12 months.
  BASDAI scale 0-10 (the higher the score the more severe the symptoms). Association between specific microbial profile and higher or lower disease activity assessed by BASDAI indicates a positive outcome.
Association between specific intestinal pathogens and disease activity as assessed by CRP concentration. | 7 stool microbial samples and 7 CRP measurements within 12 months.
  Association between specific intestinal pathogens and (higher or lower) CRP concentration compared to patients with different microbial profile indicates a positive outcome.
Association between gut wall cytokine expression and disease activity as assessed by BASDAI score. | Intestinal biopsies at baseline.
  BASDAI scale 0-10 (the higher the score the more severe the symptoms). Association between the level of cytokine expression and BASDAI score indicates a positive outcome.
Association between gut wall inflammasome activity and disease activity as assessed by BASDAI score. | Intestinal biopsies at baseline.
  BASDAI scale 0-10 (the higher the score the more severe the symptoms). Association between gut wall inflammation as assessed by inflammasome activity and disease activity as assessed by BASDAI score indicates a positive outcome.
Association between gut wall cytokine expression and disease activity as assessed by CRP concentration. | Intestinal biopsies at baseline.
  Association between gut wall inflammation as assessed by the level of cytokine expression and the disease activity as assessed by CRP concentration indicates a positive outcome.
Association between gut wall inflammasome activity and disease activity as assessed by CRP concentration. | Intestinal biopsies at baseline.
  Association between gut wall inflammation as assessed by inflammasome activity and disease activity as assessed by CRP concentration indicates a positive outcome.
Association between F-Calpro level and disease activity as assessed by BASDAI score. | 7 F-Calpro- measurements and 5 BASDAI measurements within 12 months.
  Calprotectin- level < 100 ug/l is considered as normal. BASDAI scale 0-10 (the higher the score the more severe the symptoms). Association between gut wall inflammation as assessed by F-Calpro level and disease activity as assessed by BASDAI score indicates a positive outcome.
Association between F-Calpro level and disease activity as assessed by CRP concentration. | 7 F-Calpro and CRP measurements within 12 months.
  Calprotectin- level < 100 ug/l is considered as normal. Association between gut wall inflammation as assessed by F-Calpro and disease activity as assessed by CRP concentration indicates a positive outcome.
The effect of FMT on gut wall permeability as assessed by blood zonulin concentration. | 5 measurements within 12 months.
  Change in zonulin concentration indicates a positive outcome.
The effect of FMT on gut wall bacterial penetrance as assessed by lipopolysaccharide (LPS) concentration. | 5 measurements within 12 months.
  Change in LPS concentration indicates a positive outcome.
The effect of FMT on gastrointestinal symptoms as assessed by GSRS (The Gastrointestinal Symptom Rating Scale). | 5 GSRS evaluations within 12 months.
  GSRS score scale 15-105. The higher the score the more severe the symptoms. Decrease in GSRS indicates a positive outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kari K Eklund, PhD, MD, Study Director — Hospital District of Helsinki and Uusimaa
Locations (1):
- Hospital District of Helsinki and Uusimaa, Department of Rheumatology, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Anderson JL, Edney RJ, Whelan K. Systematic review: faecal microbiota transplantation in the management of inflammatory bowel disease. Aliment Pharmacol Ther. 2012 Sep;36(6):503-16. doi: 10.1111/j.1365-2036.2012.05220.x. Epub 2012 Jul 25. PMID 22827693
- [Background] Breban M, Tap J, Leboime A, Said-Nahal R, Langella P, Chiocchia G, Furet JP, Sokol H. Faecal microbiota study reveals specific dysbiosis in spondyloarthritis. Ann Rheum Dis. 2017 Sep;76(9):1614-1622. doi: 10.1136/annrheumdis-2016-211064. Epub 2017 Jun 12. PMID 28606969
- [Background] Ciccia F, Bombardieri M, Principato A, Giardina A, Tripodo C, Porcasi R, Peralta S, Franco V, Giardina E, Craxi A, Pitzalis C, Triolo G. Overexpression of interleukin-23, but not interleukin-17, as an immunologic signature of subclinical intestinal inflammation in ankylosing spondylitis. Arthritis Rheum. 2009 Apr;60(4):955-65. doi: 10.1002/art.24389. PMID 19333939
- [Background] Ciccia F, Ferrante A, Triolo G. Intestinal dysbiosis and innate immune responses in axial spondyloarthritis. Curr Opin Rheumatol. 2016 Jul;28(4):352-8. doi: 10.1097/BOR.0000000000000296. PMID 27214393
- [Background] Ciccia F, Guggino G, Rizzo A, Alessandro R, Luchetti MM, Milling S, Saieva L, Cypers H, Stampone T, Di Benedetto P, Gabrielli A, Fasano A, Elewaut D, Triolo G. Dysbiosis and zonulin upregulation alter gut epithelial and vascular barriers in patients with ankylosing spondylitis. Ann Rheum Dis. 2017 Jun;76(6):1123-1132. doi: 10.1136/annrheumdis-2016-210000. Epub 2017 Jan 9. PMID 28069576
- [Background] Costello ME, Ciccia F, Willner D, Warrington N, Robinson PC, Gardiner B, Marshall M, Kenna TJ, Triolo G, Brown MA. Brief Report: Intestinal Dysbiosis in Ankylosing Spondylitis. Arthritis Rheumatol. 2015 Mar;67(3):686-691. doi: 10.1002/art.38967. PMID 25417597
- [Background] De Vos M, Mielants H, Cuvelier C, Elewaut A, Veys E. Long-term evolution of gut inflammation in patients with spondyloarthropathy. Gastroenterology. 1996 Jun;110(6):1696-703. doi: 10.1053/gast.1996.v110.pm8964393.
- [Background] Huttenhower C, Kostic AD, Xavier RJ. Inflammatory bowel disease as a model for translating the microbiome. Immunity. 2014 Jun 19;40(6):843-54. doi: 10.1016/j.immuni.2014.05.013. PMID 24950204
- [Background] Jalanka J, Mattila E, Jouhten H, Hartman J, de Vos WM, Arkkila P, Satokari R. Long-term effects on luminal and mucosal microbiota and commonly acquired taxa in faecal microbiota transplantation for recurrent Clostridium difficile infection. BMC Med. 2016 Oct 11;14(1):155. doi: 10.1186/s12916-016-0698-z. PMID 27724956
- [Background] Knodler LA, Crowley SM, Sham HP, Yang H, Wrande M, Ma C, Ernst RK, Steele-Mortimer O, Celli J, Vallance BA. Noncanonical inflammasome activation of caspase-4/caspase-11 mediates epithelial defenses against enteric bacterial pathogens. Cell Host Microbe. 2014 Aug 13;16(2):249-256. doi: 10.1016/j.chom.2014.07.002. PMID 25121752
- [Background] Leirisalo-Repo M, Turunen U, Stenman S, Helenius P, Seppala K. High frequency of silent inflammatory bowel disease in spondylarthropathy. Arthritis Rheum. 1994 Jan;37(1):23-31. doi: 10.1002/art.1780370105. PMID 8129761
- [Background] Mattila E, Uusitalo-Seppala R, Wuorela M, Lehtola L, Nurmi H, Ristikankare M, Moilanen V, Salminen K, Seppala M, Mattila PS, Anttila VJ, Arkkila P. Fecal transplantation, through colonoscopy, is effective therapy for recurrent Clostridium difficile infection. Gastroenterology. 2012 Mar;142(3):490-6. doi: 10.1053/j.gastro.2011.11.037. Epub 2011 Dec 7. PMID 22155369
- [Background] Nurmi K, Virkanen J, Rajamaki K, Niemi K, Kovanen PT, Eklund KK. Ethanol inhibits activation of NLRP3 and AIM2 inflammasomes in human macrophages--a novel anti-inflammatory action of alcohol. PLoS One. 2013 Nov 11;8(11):e78537. doi: 10.1371/journal.pone.0078537. eCollection 2013. PMID 24244322
- [Background] Nurmi K, Kareinen I, Virkanen J, Rajamaki K, Kouri VP, Vaali K, Levonen AL, Fyhrquist N, Matikainen S, Kovanen PT, Eklund KK. Hemin and Cobalt Protoporphyrin Inhibit NLRP3 Inflammasome Activation by Enhancing Autophagy: A Novel Mechanism of Inflammasome Regulation. J Innate Immun. 2017;9(1):65-82. doi: 10.1159/000448894. Epub 2016 Sep 22. PMID 27655219
- [Background] Rajamaki K, Lappalainen J, Oorni K, Valimaki E, Matikainen S, Kovanen PT, Eklund KK. Cholesterol crystals activate the NLRP3 inflammasome in human macrophages: a novel link between cholesterol metabolism and inflammation. PLoS One. 2010 Jul 23;5(7):e11765. doi: 10.1371/journal.pone.0011765. PMID 20668705
- [Background] Rajamaki K, Nordstrom T, Nurmi K, Akerman KE, Kovanen PT, Oorni K, Eklund KK. Extracellular acidosis is a novel danger signal alerting innate immunity via the NLRP3 inflammasome. J Biol Chem. 2013 May 10;288(19):13410-9. doi: 10.1074/jbc.M112.426254. Epub 2013 Mar 25. PMID 23530046
- [Background] Tailford LE, Crost EH, Kavanaugh D, Juge N. Mucin glycan foraging in the human gut microbiome. Front Genet. 2015 Mar 19;6:81. doi: 10.3389/fgene.2015.00081. eCollection 2015. PMID 25852737
- [Background] Taurog JD, Richardson JA, Croft JT, Simmons WA, Zhou M, Fernandez-Sueiro JL, Balish E, Hammer RE. The germfree state prevents development of gut and joint inflammatory disease in HLA-B27 transgenic rats. J Exp Med. 1994 Dec 1;180(6):2359-64. doi: 10.1084/jem.180.6.2359. PMID 7964509
- [Background] Tito RY, Cypers H, Joossens M, Varkas G, Van Praet L, Glorieus E, Van den Bosch F, De Vos M, Raes J, Elewaut D. Brief Report: Dialister as a Microbial Marker of Disease Activity in Spondyloarthritis. Arthritis Rheumatol. 2017 Jan;69(1):114-121. doi: 10.1002/art.39802. Epub 2016 Dec 1. PMID 27390077
- [Background] Van Praet L, Van den Bosch FE, Jacques P, Carron P, Jans L, Colman R, Glorieus E, Peeters H, Mielants H, De Vos M, Cuvelier C, Elewaut D. Microscopic gut inflammation in axial spondyloarthritis: a multiparametric predictive model. Ann Rheum Dis. 2013 Mar;72(3):414-7. doi: 10.1136/annrheumdis-2012-202135. Epub 2012 Nov 8. PMID 23139267
- [Derived] Parthasarathy R, Santiago F, McCluskey P, Kaakoush NO, Tedla N, Wakefield D. The microbiome in HLA-B27-associated disease: implications for acute anterior uveitis and recommendations for future studies. Trends Microbiol. 2023 Feb;31(2):142-158. doi: 10.1016/j.tim.2022.08.008. Epub 2022 Sep 1. PMID 36058784